CLINICAL TRIAL: NCT04005755
Title: A Phase 3, Open-Label, Multiple-Dose, Single-Arm Exposure Study of Maxigesic® IV in Patients With Acute Pain Following Orthopedic, General or Plastic Surgery
Brief Title: Maxigesic® IV Phase 3 Exposure Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AFT Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFT-MXIV-11
Record Dates: First submitted 2019-06-19; First posted 2019-07-02 (Actual); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain
Keywords: Analgesic
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Maxigesic® IV (Experimental): Acetaminophen 10 mg/ml + ibuprofen 3 mg/ml in 100 ml solution for infusion. The study drug will be administered by injection into a dedicated indwelling venous cannula, infused over 15 minutes. The study drug will be administered every 6 hours (q6h) for a minimum of 48 hours up to at least 5 days, with a maximum of 4 doses within a 24 hour period.
  Interventions: Drug: Maxigesic® IV

INTERVENTIONS:
Drug: Maxigesic® IV — acetaminophen 1000 mg + ibuprofen 300 mg, 100 ml solution for infusion

SUMMARY:
The study aims to determine the tolerability of repeated doses of Maxigesic® IV over an extended period of exposure.

DETAILED DESCRIPTION:
Combined administration of acetaminophen and ibuprofen has been shown to provide superior analgesia over administration of comparable doses of either component alone or placebo, when given as an intravenous formulation or as a solid oral tablet in the postoperative setting.

The superior efficacy of the combination does not appear to come at the expense of tolerability. A previous study of Maxigesic® IV in bunionectomy patients found that there were no differences between patients treated with repeated doses of Maxigesic® IV and those treated with intravenous acetaminophen, ibuprofen or placebo in the rate of discontinuations due to adverse events (AEs), the overall incidence of treatment-emergent AEs (TEAEs) or the severity of TEAEs. The incidence of common TEAEs (affecting ≥ 10% of the study population), including gastrointestinal disorders, nervous system disorders, general disorders and administration site conditions, and skin and subcutaneous tissue disorders, was not changed due to combined administration of acetaminophen and ibuprofen in Maxigesic® IV.

This study aims to determine the tolerability of repeated doses of Maxigesic® IV over an extended period of exposure (≥ 48 hours).

ELIGIBILITY:
Inclusion Criteria:

* Is male or female ≥ 18 years of age.
* Is classified by the anesthesiologist as P1 to P2 in the American Society of Anesthesiologists (ASA) Physical Status Classification System.
* Requires multiple doses of parenterally administered nonopioid analgesics over multiple days as a result of surgery (non-laparoscopic general, plastic or orthopedic surgery).
* Has an expected stay in facility ≥ 48 hours.
* Has a body weight ≥ 45 kg.
* If female and of childbearing potential, is nonlactating and nonpregnant.
* If female, is either not of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or practicing 1 of the following medically acceptable methods of birth control: i) Hormonal methods such as oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle (based on the subject's usual menstrual cycle period) before study drug administration; ii) Total abstinence from sexual intercourse since the last menses before study drug administration through completion of final study visit; iii) Intrauterine device (IUD); iv) Double-barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream).
* Is able to provide written informed consent to participate in the study and able to understand the procedures and study requirements.
* Must voluntarily sign and date an informed consent form (ICF) that is approved by an Institutional Review Board (IRB) before the conduct of any study procedure.
* Is willing and able to remain at the study site for at least 48 hours and to attend a follow-up visit at 7 ± 2 days after the last dose of study drug.

Exclusion Criteria:

* Has a known history of allergic reaction or clinically significant intolerance to acetaminophen, aspirin, opioids, or any nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen); history of NSAID-induced bronchospasm (subjects with the triad of asthma, nasal polyps, and chronic rhinitis are at greater risk for bronchospasm and should be considered carefully); or hypersensitivity, allergy, or significant reaction to sulfa (including sulfonamide) medicines, ingredients of the study drug, or any other drugs used in the study including anesthetics and antibiotics that may be required on the day of surgery.
* Has experienced any surgical complications or other issues that, in the opinion of the Investigator, could compromise the safety of the subject if he or she participates in the study or could confound the results of the study.
* Has a known or suspected history of alcoholism or drug abuse or misuse within 2 years of screening or evidence of tolerance or physical dependence before dosing with study drug.
* Has any clinically significant unstable cardiac, respiratory, neurological, immunological, hematological, or renal disease or any other condition that, in the opinion of the Investigator, could compromise the subject's welfare, ability to communicate with the study staff, or otherwise contraindicate study participation.
* Has a history or current diagnosis of a significant psychiatric disorder that, in the opinion of the Investigator, would affect the subject's ability to comply with the study requirements.
* Has tested positive either on the urine drug screen or on the alcohol breathalyzer test. Subjects who test positive and can produce a prescription for the medication from their physician may be considered for study enrolment at the discretion of the Investigator.
* Has a history of a clinically significant (Investigator opinion) gastrointestinal (GI) event within 6 months before screening or has any history of peptic or gastric ulcers or GI bleeding.
* Has a surgical or medical condition of the GI or renal system that might significantly alter the absorption, distribution, or excretion of any drug substance.
* Is considered by the Investigator, for any reason to be an unsuitable candidate to receive the study drug.
* Is receiving systemic chemotherapy, has an active malignancy of any type, or has been diagnosed with cancer within 5 years before Screening (excluding treated squamous or basal cell carcinoma of the skin).
* Is currently receiving anticoagulants (e.g. heparin or warfarin).
* Has received a course of systemic corticosteroids (either oral or parenteral) within 3 months before screening (inhaled nasal steroids and regional/limited area application of topical corticosteroids (Investigator discretion) are allowed).
* Has a history of chronic use (defined as daily use for > 2 weeks) of NSAIDs, opiates, or glucocorticoids (except inhaled nasal steroids and regional/limited topical corticosteroids), for any condition within 6 months before study drug administration. Aspirin at a daily dose of ≤ 325 mg is allowed for cardiovascular prophylaxis if the subject has been on a stable dose regimen for ≥ 30 days before screening and has not experienced any relevant medical problem.
* Has a significant renal or hepatic disease, as indicated by clinical laboratory assessment (results ≥ 3 times the upper limit of normal [ULN] for any liver function test, including aspartate aminotransferase [AST], alanine aminotransferase [ALT], or creatinine ≥ 1.5 times the ULN).
* Has any clinically significant laboratory finding at screening that, in the opinion of the Investigator, contraindicates study participation.
* Previously participated in another clinical study of Maxigesic® IV or received any investigational drug or device or investigational therapy within 30 days before Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Gottlieb, DPM, Principal Investigator — Chesapeake Research Group; Simon Carson, MD, Principal Investigator — Southern Clinical Trials Ltd; Gregory L Ruff, MD, Principal Investigator — Chapel Hill Research Group; Nigel Gilchrist, MD, Principal Investigator — CGM Research Trust
Locations (4):
- United States (2):
  - Chesapeake Reserach Group, Pasadena, Maryland
  - Chapel Hill Research Group, Chapel Hill, North Carolina
- New Zealand (2):
  - Canterbury Geriatric Medical Research Trust, Christchurch
  - Southern Clinical Trials, Christchurch

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 323 subjects were screened, of whom 90 subjects were screening failures, and a total of 233 subjects were enrolled. 1 subject was enrolled but not dosed due to receiving prohibited concomitant medications during surgery, therefore a total of 232 subjects were administered at least one dose of the study drug. 17 subjects discontinued from the study, including 14 discontinuations during the treatment period, and 3 discontinuations during the follow-up period. 215 subjects completed the full study
Period: Overall Study
Arm/Group | Maxigesic® IV
Started | 232
Completed | 215
Not Completed | 17
Not completed — Adverse Event | 6
Not completed — Physician Decision | 3
Not completed — Administrative reason, temporary site closure due to COVID-19 | 4
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 171
  >=65 years | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144
  Male | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 223
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 91
  White | 131
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 85
  United States | 147
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of TEAEs (Treatment-emergent Adverse Events)
Description: The incidence of treatment-emergent adverse events associated with exposure Maxigesic® IV
Time Frame: During treatment period (≥ 48 hours - 5 days)
Population: The safety analysis was on all participants who were administered at least one dose of study medication, with treatment allocation for analysis based on the actual treatment the participant received.
Measure: Number; unit: Treatment-Emergent Adverse Events
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
Treatment-Emergent Adverse Events
  Incidence of TEAEs ( 2 days treatment): number analyzed (Participants) | 182
  Incidence of TEAEs ( 2 days treatment) | 256
  Incidence of TEAEs (5 days treatment): number analyzed (Participants) | 50
  Incidence of TEAEs (5 days treatment) | 38

2. Secondary Outcome: Time Course of TEAEs
Description: The incidence of treatment-emergent adverse events associated with exposure Maxigesic® IV during various study time periods
Time Frame: After receiving the first dose of study medication until 7 days after the last dose, a total of approximately 9 days for subjects who received the treatment for 48 hours and 12 days for subjects who received the treatment for 5 days.
Population: as for outcome 1
Measure: Number; unit: Treatment-Emergent Adverse Events
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
Treatment-Emergent Adverse Events
  Treatment-Emergent Adverse Events Day 1 | 166
  Treatment-Emergent Adverse Events Day 2: number analyzed (Participants) | 224
  Treatment-Emergent Adverse Events Day 2 | 90
  Treatment-Emergent Adverse Events Day 3: number analyzed (Participants) | 52
  Treatment-Emergent Adverse Events Day 3 | 9
  Treatment-Emergent Adverse Events Day 4: number analyzed (Participants) | 50
  Treatment-Emergent Adverse Events Day 4 | 12
  Treatment-Emergent Adverse Events Day 5: number analyzed (Participants) | 50
  Treatment-Emergent Adverse Events Day 5 | 17

3. Secondary Outcome: Incidence of TRAEs (Treatment-related Adverse Events)
Description: The incidence of treatment-related adverse events (TEAEs considered by the investigator to be "probably" or "definitely" related to the study drug) associated with exposure Maxigesic® IV
Time Frame: During treatment period (≥ 48 hours - 5 days)
Population: as for outcome 1
Measure: Number; unit: Treatment-Emergent Adverse Events
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
Treatment-Emergent Adverse Events
  Not related | 103
  Unlikely | 89
  Possible | 34
  Probable | 17
  Definite | 51

4. Secondary Outcome: Incidence of TEAEs of Interest
Description: The incidence of TEAEs of interest (cardiovascular, gastrointestinal, renal, hepatic, administration site conditions and bleeding-related events)
Time Frame: During treatment period (≥ 48 hours - 5 days)
Population: as for outcome 1
Measure: Number; unit: Treatment-Emergent Adverse Events
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
Treatment-Emergent Adverse Events
  Gastrointestinal disorders | 67
  Renal and urinary disorders | 12
  Abnormal hepatic function lab results | 25
  General disorders and administration site conditions | 78
  Cardiac Disorders | 3
  Vascular disorders | 7

5. Secondary Outcome: Changes in Blood Pressure
Description: Systolic and Diastolic Blood Pressured Measured every 24 hours
Time Frame: From the baseline (Day 1 prior to surgery) until 7 days after the last dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
mmHg
  Systolic Blood Pressure change from the baseline | -0.9 (18.98)
  Diastolic Blood Pressure change from the baseline | -0.5 (11.31)

6. Secondary Outcome: Changes in Heart Rate
Description: Measured every 24 hours
Time Frame: From the baseline (Day 1 prior to surgery) until 7 days after the last dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
beats/min | 3.4 (11.86)

7. Secondary Outcome: Changes in Temperature
Description: Measured every 24 hours
Time Frame: From the baseline (Day 1 prior to surgery) until 7 days after the last dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
degree Celsius | 0.2 (0.38)

8. Secondary Outcome: Changes in Respiratory Rate
Description: Respiratory Rate Measured every 24 hours
Time Frame: From the baseline (Day 1 prior to surgery) until 7 days after the last dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
breaths/min | 0.5 (2.43)

9. Secondary Outcome: Changes in Hematology Values (Hemoglobin)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
g/L | -11.6 (13.4)

10. Secondary Outcome: Changes in Hematology Values (Hematocrit)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of red blood cells in blood
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
proportion of red blood cells in blood | -0.03 (0.04)

11. Secondary Outcome: Changes in Hematology Values (Platelet Count)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: billions/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
billions/L | -12.8 (40.1)

12. Secondary Outcome: Changes in Hematology Values (Red Blood Cell Count)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: trillions/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
trillions/L | -0.4 (0.5)

13. Secondary Outcome: Changes in Hematology Values (White Blood Cell Count)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: billions/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
billions/L | 6.2 (1.7)

14. Secondary Outcome: Changes in Hematology Values (Differential Leukocyte Count)
Description: Hematology test was Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: billions/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
billions/L
  Basophils | -0.00 (0.02)
  Eosinophils | 0.05 (0.13)
  Lymphocytes | -0.2 (0.5)
  Monocytes | 0.2 (0.2)
  Neutrophils | 1.5 (1.7)

15. Secondary Outcome: Changes in Blood Biochemistry Values (Sodium)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
mmol/L | -0.6 (2.3)

16. Secondary Outcome: Changes in Blood Biochemistry Values (Potassium)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
mmol/L | -0.1 (0.4)

17. Secondary Outcome: Changes in Blood Biochemistry Values (Urea)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
mmol/L | -0.7 (1.4)

18. Secondary Outcome: Changes in Blood Biochemistry Values (Creatinine)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
μmol/L | -3.9 (9.5)

19. Secondary Outcome: Changes in Blood Biochemistry Values (Phosphate)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
mmol/L | -0.1 (0.2)

20. Secondary Outcome: Changes in Blood Biochemistry Values (Glucose)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
mmol/L | 0.7 (1.5)

21. Secondary Outcome: Changes in Blood Biochemistry Values (Albumin)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
g/L | -4.9 (3.2)

22. Secondary Outcome: Changes in Blood Biochemistry Values (Total Protein)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
g/L | -5.8 (5.3)

23. Secondary Outcome: Changes in Blood Biochemistry Values (Alkaline Phosphates)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
IU/L | -2.1 (15.1)

24. Secondary Outcome: Changes in Blood Biochemistry Values (Gamma-glutamyl Transferase)
Description: Blood Biochemistry was Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
IU/L | 4.3 (16.5)

25. Secondary Outcome: Changes in Blood Biochemistry Values (Aspartate Transaminase)
Description: Blood Chemistry (AST) was Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
IU/L | 7.1 (23.3)

26. Secondary Outcome: Changes in Blood Biochemistry Values (Alanine Transaminase)
Description: Blood Chemistry (ALT) was Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
IU/L | 4.5 (25.2)

27. Secondary Outcome: Changes in Blood Biochemistry Values (Bilirubin)
Description: Measured at screening visit and at the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
μmol/L | 0.0 (3.9)

28. Secondary Outcome: Changes in ECG (Electrocardiography) Status (Normal/Abnormal)
Description: All components of the ECG will be analysed to assess safety (P wave, QRS Complex, QT interval, PR interval, T wave, ST segment, U wave, PR segment) in 5 categories of the shift from baseline to the end of treatment from:
  Normal to Normal Normal to Abnormal NCS (Non-clinically Significant) Abnormal NCS to Normal Abnormal NCS to Abnormal NCS Missing
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
Participants
  Shift from Baseline to the end of treatment Missing | 2
  Shift from Baseline to the end of treatment Normal to Normal | 83
  Shift from Baseline to the end of treatment Normal to Abnormal NCS | 18
  Shift from Baseline to the end of treatment Abnormal NCS to Normal | 44
  Shift from Baseline to the end of treatment Abnormal NCS to Abnormal NCS | 85

29. Secondary Outcome: Changes in Hepatic Enzymes From Baseline to the End of the Treatment
Description: The elevation in hepatic enzymes (ALP, ALT, AST, GGT) from baseline to the end of the treatment
Time Frame: Prior to surgery, on Day 1 and at discharge (Day 5)
Population: The safety analysis was on all participants who were administered at least one dose of study medication, with treatment allocation for analysis based on the actual treatment the participant received. The number of participants analyzed are reporting the number of participants who experienced the shifts from Normal to Abnormal.
Measure: Count of Participants; unit: Participants
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
Participants
  Shifts from Normal to High Upper Limit of Normal (ULN) <3.0: number analyzed (Participants) | 59
  Shifts from Normal to High Upper Limit of Normal (ULN) <3.0: ALP | 1
  Shifts from Normal to High Upper Limit of Normal (ULN) <3.0: ALT | 24
  Shifts from Normal to High Upper Limit of Normal (ULN) <3.0: AST | 22
  Shifts from Normal to High Upper Limit of Normal (ULN) <3.0: GGT | 12
  Shift from Normal to High ULN ≥ 3.0, <5.0: number analyzed (Participants) | 9
  Shift from Normal to High ULN ≥ 3.0, <5.0: ALP | 0
  Shift from Normal to High ULN ≥ 3.0, <5.0: ALT | 4
  Shift from Normal to High ULN ≥ 3.0, <5.0: AST | 5
  Shift from Normal to High ULN ≥ 3.0, <5.0: GGT | 0
  Shift from Normal to High ULN ≥ 5.0: number analyzed (Participants) | 2
  Shift from Normal to High ULN ≥ 5.0: ALP | 0
  Shift from Normal to High ULN ≥ 5.0: ALT | 2
  Shift from Normal to High ULN ≥ 5.0: AST | 0
  Shift from Normal to High ULN ≥ 5.0: GGT | 0

30. Secondary Outcome: Patient's Global Evaluation of the Study Drug
Description: Summary of the patients' ratings of the study medication (1 = Poor; 2 = Fair; 3 = Good; 4 = Very Good; 5 = Excellent)
Time Frame: 5 days after the first dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Maxigesic® IV
Number analyzed (Participants) | 232
Participants
  Poor | 4
  Fair | 12
  Good | 40
  Very Good | 82
  Excellent | 93
  Missing | 1

ADVERSE EVENTS:
Time Frame: During the treatment period (after receiving the first dose of study medication until 7 days after the last dose, a total of approximately 12 days)
Description: Treatment-emergent adverse events (TEAEs): Treatment-emergent adverse events (TEAEs) were defined as events that emerged during treatment, having been absent pre-treatment, or that worsened relative to the pre-treatment status.
  The definition of serious adverse events and reporting requirement are determined in the study protocol section 8.1.2 and section 8.4
Arm/Group | Maxigesic® IV
All-Cause Mortality (participants affected / at risk) | 0/232
Serious Adverse Events (participants affected / at risk) | 2/232
Other Adverse Events (participants affected / at risk) | 164/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maxigesic® IV (N=232)
hypotension (Vascular disorders) | 1 (1) — The subject experienced hypotension (primary event) resulting in hospitalization after receiving the second dose of study medication. blood pressure: 67/49mmHg. The SAE was evaluated as "unlikely related to the investigational product.
bowel obstruction (Gastrointestinal disorders) | 1 (1) — the subject developed symptoms of bowel obstruction with nausea, vomiting with abdomen distended 3 days after the surgery and resulted in hospitalization. The SAE was evaluated as "unlikely related to the investigational product"
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maxigesic® IV (N=232)
Infusion site pain (General disorders) | 44 (49) — Infusion site pain
Nausea (Gastrointestinal disorders) | 28 (32) — Nausea
Infusion site extravasation (General disorders) | 18 (19) — Infusion site extravasation
Constipation (Gastrointestinal disorders) | 18 (19) — Constipation
Headache (Nervous system disorders) | 13 (13) — Headache
Dizziness (Nervous system disorders) | 9 (12) — Dizziness
Polyuria (Renal and urinary disorders) | 9 (9) — Polyuria
Procedural nausea (Injury, poisoning and procedural complications) | 8 (8) — Procedural nausea
Somnolence (Nervous system disorders) | 7 (7) — Somnolence
Diarrhoea (Nervous system disorders) | 5 (5) — Diarrhoea
Alanine aminotransferase increased (Hepatobiliary disorders) | 5 (5) — Alanine aminotransferase increased

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT04005755/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT04005755/SAP_001.pdf